CLINICAL TRIAL: NCT03530800
Title: A Double-Blind, Placebo-Controlled Study of Dronabinol in Trichotillomania and Other Body Focused Repetitive Behaviors
Brief Title: Dronabinol in Trichotillomania and Other Body Focused Repetitive Behaviors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB18-0542
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Trichotillomania; Skin-Picking
MeSH Terms: conditions — Trichotillomania; Excoriation Disorder | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dronabinol (Active Comparator): Subjects will receive dronabinol 5mg once daily for two weeks, 5mg twice daily for the subsequent two weeks, and 5mg three times daily for the final six weeks. Dose escalations will only be done if the investigator deems necessary.
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): Subjects will receive placebo for 10 weeks weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol for 10 weeks (5mg per day first 2 weeks, 10mg per day second two weeks, 15mg per day last six weeks)
  Other Names: Marinol
  Arms: Dronabinol
Drug: Placebo — Placebo for 10 weeks
  Arms: Placebo

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of dronabinol in trichotillomania and other body-focused repetitive behaviors such as skin-picking disorder. 50 subjects with DSM-5 trichotillomania or skin-picking disorder will receive 10 weeks of double-blind dronabinol or placebo. The hypothesis to be tested is that dronabinol will be effective and well tolerated in patients with trichotillomania and/or skin-picking disorder compared to placebo. The proposed study will provide needed data on the treatment of disabling disorders that currently lacks a clearly effective treatment.

DETAILED DESCRIPTION:
Pathological hair-pulling, trichotillomania, has been defined as repetitive, intentionally performed pulling that causes noticeable hair loss and results in clinically significant distress or functional impairment. Although discussed in the medical literature for over one hundred years, and affecting all strata of society, there have been no epidemiological studies detailing how common trichotillomania is and there are no clear treatment approaches for everyone with trichotillomania. Behavioral therapy is generally regarded as the first-line treatment but trained therapists are difficult to find. In addition, there is no medication currently approved by the Food and Drug Administration for trichotillomania. Trichotillomania is related clinically to other BFRBs, specifically skin picking disorder. In fact, it appears that trichotillomania and skin picking disorder may in fact share a common neurobiology. Other BFRBs such as skin ppicking disorder also lack any agreed upon medication intervention, but evidence suggests that both skin picking disorder and trichotillomania may respond to the same interventions.

The Trichotillomania Impact Project survey showed that only 15% of adults in the community with trichotillomania reported experiencing significant improvement with treatment of their symptoms. This may be because of the ongoing difficulty of finding a therapist experienced in trichotillomania treatments. More than 55% of persons in this survey believed that their clinician did not have sufficient knowledge of the disorder, and less than one-third were receiving evidence-based treatments for trichotillomania.

A recent meta-analytic study of randomized treatment trials in adults demonstrated that behavioral treatments, mainly habit reversal therapy, have the greatest efficacy in treatment of trichotillomania. Selective serotonin reuptake inhibitors (SSRIs) are the most widely used treatment for adults with trichotillomania, despite evidence that their efficacy is no greater than placebo.

Instead of using SSRIs, the investigators conducted an open-label study of dronabinol a synthetic form of tetrahydrocannabinol (THC) approved by the FDA as an appetite stimulant for people with AIDS and antiemetic for people receiving chemotherapy, in 14 women with trichotillomania and found that 9 (64.3%) responded to treatment and that the mean effective dose was 11.6 ± 4.1 mg/day.

A recent study using diffusion tensor imaging demonstrated that both trichotillomania and skin-picking subjects exhibited significantly reduced fractional anisotropy in anterior cingulate, presupplementary motor area, and temporal cortices. These data suggest that the disorganization of white matter tracts in motor habit generation and suppression may underlie the pathophysiology of these disorders. Neurochemically, motor habits may rely partially on the endocannabinoid system. CB1 receptors are highly expressed in the basal ganglia nuclei, the hippocampus, cerebellum, and neocortex and are implicated in attenuating glutamatergic exocitotoxic damage by suppressing the neuronal release of glutamate via inhibition of calcium channels. The activation of CB1 receptors reduces glutamate release in the dorsal and ventral striatum [possibly through an interaction with brain-derived neurotrophic factor], thereby modulating neurotransmission in the basal ganglia and mesolimbic reward system . Stress-induced anxious behavior has been associated with the loss of CB1 receptor function in the striatum.

Glutamatergic dysfunction has been implicated in the pathophysiology of trichotillomania. Pharmacotherapies, such as dronabinol, that target excessive glutamatergic drive through its effects on CB! Receptors may, therefore, be expected to correct the underlying pathophysiology and symptoms of trichotillomania.

In the USA, dronabinol is FDA-approved for the treatment of anorexia associated with weight loss in patients with AIDS and nausea and vomiting associated with cancer chemotherapy. In our previous study examining dronabinol for trichotillomania, doses between 5 and 15mg/day were well tolerated and beneficial. This lack of significant side effects is consistent with other studies of dronabinol where it has been associated primarily with central nervous system-related adverse events (for example, confusion, dizziness, euphoria, and somnolence), but these adverse events are generally mild to moderate in severity and generally reversible upon dose modification.

Given the serious personal consequences associated with trichotillomania, and the likelihood of success of dronabinol in treating the disorder, the aim of the present study was to examine the efficacy and safety of dronabinol vs placebo in adults with trichotillomania using a double-blind, placebo-controlled design.

The investigators hypothesize that dronabinol will be more effective than placebo in reducing the frequency of hair pulling and in improving overall psychosocial functioning after 10 weeks of treatment when compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* current DSM-5 trichotillomania
* ability to understand and sign the consent form

Exclusion Criteria:

* Unstable Medical illness based on history of clinically significant abnormalities on baseline physical examination
* Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
* Subjects considered an immediate suicide risk based on the Columbia Suicide Severity Rating Scale (C-SSRS) (www.cssrs.columbia.edu/docs)
* Past 12-month DSM-5 psychiatric disorder other than trichotillomania
* Illegal substance use based on urine toxicology screening
* Use of any other psychotropic medication (except a PRN hypnotic)
* Previous treatment with dronabinol
* Cognitive impairment that interferes with the capacity to understand and self administer medication or provide written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Woods DW, Flessner CA, Franklin ME, Keuthen NJ, Goodwin RD, Stein DJ, Walther MR; Trichotillomania Learning Center-Scientific Advisory Board. The Trichotillomania Impact Project (TIP): exploring phenomenology, functional impairment, and treatment utilization. J Clin Psychiatry. 2006 Dec;67(12):1877-88. doi: 10.4088/jcp.v67n1207. PMID 17194265
- [Background] Bloch MH, Landeros-Weisenberger A, Dombrowski P, Kelmendi B, Wegner R, Nudel J, Pittenger C, Leckman JF, Coric V. Systematic review: pharmacological and behavioral treatment for trichotillomania. Biol Psychiatry. 2007 Oct 15;62(8):839-46. doi: 10.1016/j.biopsych.2007.05.019. Epub 2007 Aug 28. PMID 17727824
- [Background] Grant JE, Odlaug BL, Chamberlain SR, Kim SW. Dronabinol, a cannabinoid agonist, reduces hair pulling in trichotillomania: a pilot study. Psychopharmacology (Berl). 2011 Dec;218(3):493-502. doi: 10.1007/s00213-011-2347-8. Epub 2011 May 19. PMID 21590520
- [Background] Chamberlain SR, Hampshire A, Menzies LA, Garyfallidis E, Grant JE, Odlaug BL, Craig K, Fineberg N, Sahakian BJ. Reduced brain white matter integrity in trichotillomania: a diffusion tensor imaging study. Arch Gen Psychiatry. 2010 Sep;67(9):965-71. doi: 10.1001/archgenpsychiatry.2010.109. PMID 20819990
- [Background] Herkenham M, Lynn AB, Little MD, Johnson MR, Melvin LS, de Costa BR, Rice KC. Cannabinoid receptor localization in brain. Proc Natl Acad Sci U S A. 1990 Mar;87(5):1932-6. doi: 10.1073/pnas.87.5.1932. PMID 2308954
- [Background] Glass M, Felder CC. Concurrent stimulation of cannabinoid CB1 and dopamine D2 receptors augments cAMP accumulation in striatal neurons: evidence for a Gs linkage to the CB1 receptor. J Neurosci. 1997 Jul 15;17(14):5327-33. doi: 10.1523/JNEUROSCI.17-14-05327.1997. PMID 9204917
- [Background] Gerdeman GL, Ronesi J, Lovinger DM. Postsynaptic endocannabinoid release is critical to long-term depression in the striatum. Nat Neurosci. 2002 May;5(5):446-51. doi: 10.1038/nn832. PMID 11976704
- [Background] Marsicano G, Goodenough S, Monory K, Hermann H, Eder M, Cannich A, Azad SC, Cascio MG, Gutierrez SO, van der Stelt M, Lopez-Rodriguez ML, Casanova E, Schutz G, Zieglgansberger W, Di Marzo V, Behl C, Lutz B. CB1 cannabinoid receptors and on-demand defense against excitotoxicity. Science. 2003 Oct 3;302(5642):84-8. doi: 10.1126/science.1088208. PMID 14526074
- [Background] Khaspekov LG, Brenz Verca MS, Frumkina LE, Hermann H, Marsicano G, Lutz B. Involvement of brain-derived neurotrophic factor in cannabinoid receptor-dependent protection against excitotoxicity. Eur J Neurosci. 2004 Apr;19(7):1691-8. doi: 10.1111/j.1460-9568.2004.03285.x. PMID 15078543
- [Background] De Chiara V, Angelucci F, Rossi S, Musella A, Cavasinni F, Cantarella C, Mataluni G, Sacchetti L, Napolitano F, Castelli M, Caltagirone C, Bernardi G, Maccarrone M, Usiello A, Centonze D. Brain-derived neurotrophic factor controls cannabinoid CB1 receptor function in the striatum. J Neurosci. 2010 Jun 16;30(24):8127-37. doi: 10.1523/JNEUROSCI.1683-10.2010. PMID 20554863
- [Background] van der Stelt M, Di Marzo V. Cannabinoid receptors and their role in neuroprotection. Neuromolecular Med. 2005;7(1-2):37-50. doi: 10.1385/NMM:7:1-2:037. PMID 16052037
- [Background] Rossi S, De Chiara V, Musella A, Kusayanagi H, Mataluni G, Bernardi G, Usiello A, Centonze D. Chronic psychoemotional stress impairs cannabinoid-receptor-mediated control of GABA transmission in the striatum. J Neurosci. 2008 Jul 16;28(29):7284-92. doi: 10.1523/JNEUROSCI.5346-07.2008. PMID 18632932
- [Background] Grant JE, Odlaug BL, Kim SW. N-acetylcysteine, a glutamate modulator, in the treatment of trichotillomania: a double-blind, placebo-controlled study. Arch Gen Psychiatry. 2009 Jul;66(7):756-63. doi: 10.1001/archgenpsychiatry.2009.60. PMID 19581567
- [Background] Bienvenu OJ, Wang Y, Shugart YY, Welch JM, Grados MA, Fyer AJ, Rauch SL, McCracken JT, Rasmussen SA, Murphy DL, Cullen B, Valle D, Hoehn-Saric R, Greenberg BD, Pinto A, Knowles JA, Piacentini J, Pauls DL, Liang KY, Willour VL, Riddle M, Samuels JF, Feng G, Nestadt G. Sapap3 and pathological grooming in humans: Results from the OCD collaborative genetics study. Am J Med Genet B Neuropsychiatr Genet. 2009 Jul 5;150B(5):710-20. doi: 10.1002/ajmg.b.30897. PMID 19051237
- [Background] Beal JE, Olson R, Laubenstein L, Morales JO, Bellman P, Yangco B, Lefkowitz L, Plasse TF, Shepard KV. Dronabinol as a treatment for anorexia associated with weight loss in patients with AIDS. J Pain Symptom Manage. 1995 Feb;10(2):89-97. doi: 10.1016/0885-3924(94)00117-4. PMID 7730690
- [Background] Beal JE, Olson R, Lefkowitz L, Laubenstein L, Bellman P, Yangco B, Morales JO, Murphy R, Powderly W, Plasse TF, Mosdell KW, Shepard KV. Long-term efficacy and safety of dronabinol for acquired immunodeficiency syndrome-associated anorexia. J Pain Symptom Manage. 1997 Jul;14(1):7-14. doi: 10.1016/S0885-3924(97)00038-9. PMID 9223837
- [Background] Swedo SE, Leonard HL, Rapoport JL, Lenane MC, Goldberger EL, Cheslow DL. A double-blind comparison of clomipramine and desipramine in the treatment of trichotillomania (hair pulling). N Engl J Med. 1989 Aug 24;321(8):497-501. doi: 10.1056/NEJM198908243210803. PMID 2761586
- [Background] Keuthen NJ, O'Sullivan RL, Ricciardi JN, Shera D, Savage CR, Borgmann AS, Jenike MA, Baer L. The Massachusetts General Hospital (MGH) Hairpulling Scale: 1. development and factor analyses. Psychother Psychosom. 1995;64(3-4):141-5. doi: 10.1159/000289003. PMID 8657844
- [Background] Grant JE, Chamberlain SR. Clinical correlates of symptom severity in skin picking disorder. Compr Psychiatry. 2017 Oct;78:25-30. doi: 10.1016/j.comppsych.2017.07.001. Epub 2017 Jul 8. PMID 28779593
- [Derived] Grant JE, Valle S, Chesivoir E, Ehsan D. Tetrahydrocannabinol fails to reduce hair pulling or skin picking: results of a double-blind, placebo-controlled study of dronabinol. Int Clin Psychopharmacol. 2022 Jan 1;37(1):14-20. doi: 10.1097/YIC.0000000000000382. PMID 34825898
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dronabinol | Placebo
Started | 25 | 25
Completed | 14 | 16
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.04 (12.48) | 28.36 (7.27) | 30.7 (10.38)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 6 | 3 | 9
  Other | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 23 | 42
  Black | 3 | 1 | 4
  Asian | 2 | 1 | 3
  Mixed | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 25 | 50
Any Psychiatric Diagnosis [Count of Participants; unit: Participants] | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: NIMH Trichotillomania Symptom Severity Scale (NIMH-TSS)
Description: The entire study lasts 10 weeks. Every two weeks subjects will take the NIMH-TSS. The change in scores from baseline to after 10 weeks will be assessed. The scale itself assesses severity of trichotillomania symptoms. The NIMH-TSS score ranges from 0 to 20, with 0 being no symptoms and 20 being the most severe.
Time Frame: Assessed every two weeks up to 10 weeks, baseline data reported
Population: Data provided for subjects that reported data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 13 | 16
score on a scale | 12.38 (3.15) | 10.63 (3.42)

2. Primary Outcome: Skin Picking Symptom Assessment Scale (SP-SAS)
Description: The entire study lasts 10 weeks. Every two weeks subjects will take the SP-SAS. The change in scores from baseline to after 10 weeks will be assessed. The scale itself assesses severity of skin-picking symptoms. The SP-SAS score ranges from 0 to 48, with 0 being no symptoms and 48 being the most severe.
Time Frame: Assessed every two weeks up to 10 weeks, baseline reported
Population: Data provided for subjects that reported data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dronabinol | Placebo
Number analyzed (Participants) | 8 | 6
score on a scale | 24.44 (9.46) | 28.5 (4.23)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the entire duration of the study (10 weeks). Subjects were asked about adverse events at each study visit and asked to reach out in between visits as well if needed to report adverse events.
Description: Definition does not differ from clinicaltrials.gov definition.
Arm/Group | Dronabinol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 16/25 | 7/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dronabinol (N=25) | Placebo (N=25)
Light headed/dizzy (General disorders) | 5 (5) | 1/1 (1)
High (easy laughing, elation, heightened awareness) (General disorders) | 4 (4) | 0 (0)
Cognitive blunting, attentional problems (Psychiatric disorders) | 4 (4) | 2 (2)
Sedation (General disorders) | 5 (5) | 3 (3)
Dry mouth (General disorders) | 4 (4) | 2 (2)
Headache (General disorders) | 0 (0) | 1 (1)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Sleep disturbance (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT03530800/Prot_SAP_001.pdf